CLINICAL TRIAL: NCT06456593
Title: A Phase 2b, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Obefazimod in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Efficacy and Safety of Obefazimod in Subjects With Moderately to Severely Active Crohn's Disease
Acronym: ENHANCE-CD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-202
Record Dates: First submitted 2024-05-16; First posted 2024-06-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Moderately to Severely Active Crohn Disease
Keywords: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Obefazimod 50mg (Experimental): Obefazimod 50mg given once-daily (QD) in subjects with moderately to severely active Crohn's disease (CD)
  Interventions: Drug: Obefazimod
- Obefazimod 25mg (Experimental): Obefazimod 25mg given once-daily (QD) in subjects with moderately to severely active Crohn's disease (CD)
  Interventions: Drug: Obefazimod
- Obefazimod 12.5mg (Experimental): Obefazimod 12.5mg given once-daily (QD) in subjects with moderately to severely active Crohn's disease (CD)
  Interventions: Drug: Obefazimod
- Placebo (Placebo Comparator): Placebo given once-daily (QD) in subjects with moderately to severely active Crohn's disease (CD)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Obefazimod — Obefazimod is administered once-daily in fed condition (ideally at the same time in the morning).
  Arms: Obefazimod 12.5mg; Obefazimod 25mg; Obefazimod 50mg
Other: Placebo — Matching placebo will be administered QD in fed condition (ideally at the same time in the morning).
  Arms: Placebo

SUMMARY:
This study has 3 treatment phases, a 12-Week Induction Phase, a 40-Week Maintenance Phase, and a 48-Week Extension Phase.

The objective is to evaluate the efficacy and safety of obefazimod compared to placebo as induction and maintenance therapy in subjects with moderately to severely active CD after inadequate response (no response, loss of response, or intolerance) to conventional therapies and/or advanced therapies.

The primary objective for the 48-Week Extension Phase is to evaluate the safety and tolerability of obefazimod compared with placebo in subjects who are enrolled in the Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (at birth) 18 to 75 years old and able to understand, sign, and date the written voluntary informed consent at the visit prior to any protocol-specified procedures
2. Able and willing to comply with study visits and procedures as per protocol.
3. Confirmed and documented diagnosis of CD based on endoscopy and histology reports.
4. Moderately to severely active CD as defined by 220 ≤ CDAI ≤ 450 and SES-CD ≥ 6 for ileo-colonic or colonic disease or SES-CD ≥ 4 for isolated ileal disease (per central reading).
5. Documented inadequate response (defined as lack of response or loss of response or intolerance) to at least one of the following treatments: corticosteroids (CS), immunosuppressants (IS), biologic or biosimilar therapies, or janus kinase (JAK) (note: failure to only 5-aminosalicylic acid [5-ASA] is not accepted)
6. Women of childbearing potential (WOCBP) and male subjects with WOCBP partner must agree to comply with contraception requirements as stated in section 4.5 (contraception) of this protocol.
7. Subject should be affiliated to a health insurance policy whenever required by a participating country or state.
8. Subject is able and willing to comply with usual public recommendations for sun protection.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will be excluded from the study:

1. WOCBP subject who is pregnant or breast-feeding at screening, or intends to become pregnant during the study; or male subject with WOCBP partner who intends to be pregnant during the study.
2. Current diagnosis of ulcerative colitis (UC) or indeterminate colitis
3. CD without ileal and/or colonic involvement
4. Untreated active external or perianal fistula or abscess. Stable fistula without abscess and with minimal or low drainage may be enrolled. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks before screening colonoscopy or 8 weeks before screening colonoscopy for intra-abdominal abscesses, if no additional surgery is anticipated.
5. Symptomatic bowel stricture and/or stenosis not passable in endoscopy
6. Related to CD surgery:

   1. Current stoma or ileoanal pouch
   2. More than 2 missing complete segments of the following 5 segments: terminal ileum, right colon, transverse colon, left colon, and sigmoid and rectum
   3. Combined previous small bowel resections > 100 cm
   4. Surgical bowel resection within the past 3 months prior to baseline
   5. Any other manifestation that might require surgery while enrolled in the study
7. Related to CD treatments:

   1. Subject who is currently treated with prohibited concomitant therapies for CD as described in the study protocol
   2. Subject who has previously received natalizumab (or any other α4β1 integrin agonist)
   3. Subject who has failed more than three advanced therapies for the treatment of CD, or two different mechanisms of action for advanced therapies of CD
8. History of, or active, malignancy including nonmelanoma skin cancer (subjects with a 5-year disease-free survival are eligible)
9. History of colonic cancer or colonic low grade or high grade dysplasia adenomatous polyps, and/or at the screening endoscopy, evidence of low grade or high grade dysplasia adenomatous polyps (fully removed or not)
10. Subject with history of, or diagnosed with, the following during screening: primary sclerosing cholangitis, autoimmune hepatitis, or primary biliary cirrhosis
11. Serious illness requiring hospitalization (not related to CD) within 4 weeks prior to screening
12. Subject with the following infectious conditions:

    1. Chronic or recurrent Grade 3 or Grade 4 infection within the last 2 months prior to screening or history of opportunistic infection while not on immunosuppressive therapy
    2. Herpes zoster reactivation within the last 2 months prior to screening
    3. Active infection at screening or any major episode of infection that required hospitalization or treatment with IV antibiotics within 1 month of screening or during screening (fungal infection of nail beds is allowed)
    4. Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) that required treatment per local medical practice or positive test for Clostridioides difficile (C. difficile) toxin at screening.
    5. Subject with human immunodeficiency virus (HIV) infection
    6. Acute or chronic hepatitis B infection at screening (positive for hepatitis B surface antigen [HbsAg] or negative for HbsAg and positive for anti-hepatitis B core antibody in conjunction with detectable hepatitis B virus [HBV] deoxyribonucleic acid [DNA], or detectable HBV DNA).
    7. Acute or chronic hepatitis C virus (HCV) infection as defined by positive for hepatitis C antibody (subjects successfully treated and without recurrence ≥ 1 year with no detectable HCV RNA [assessed centrally] are eligible)
    8. Active tuberculosis (TB) or untreated latent TB (For subjects with positive or intermediate QuantiFERON test)
13. Subject with uncontrolled ischemic heart disease and/or a history of congestive heart failure
14. Subject with a known family or personal history of congenital or acquired long QT syndrome, or subjects with a marked baseline prolongation of QT/ heart rate-corrected QT (QTc) interval
15. Subject with a history of torsade de pointe (TdP)
16. Acute or chronic clinically relevant pulmonary, hepatic, or renal functional abnormality, encephalopathy, neuropathy or unstable central nervous system pathology such as seizure disorder, or any other clinically significant medical problems.
17. Subjects who received live vaccine within 3 months prior to screening and/or subject who is planning to receive such a vaccine during the study duration
18. Acute or chronic pancreatitis
19. Subject with the following hematological and biochemical laboratory parameters obtained during the screening period:

    1. Hemoglobin ≤ 8.0 g/dL1
    2. Absolute neutrophil count < 750/mm3
    3. Platelets < 100,000 /mm3
    4. eGFR < 60 mL/min/1.73 m2
    5. Total serum bilirubin > 1.5 x ULN (except if related to pre-existing and documented Gilbert syndrome)
    6. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2 x ULN
20. Subject who does not meet the washout period requirements prior to the screening endoscopy as described in the prohibited medication section of the study protocol
21. Use of any investigational or nonregistered product within 3 months or within 5 halflives preceding baseline, whichever is longer, and during the study.
22. Subjects previously treated with obefazimod or with a known hypersensitivity to the active substance or to any of the excipients
23. Illicit drug or alcohol abuse or dependence
24. Subject who is committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
25. Any condition, which in the opinion of the investigator, could compromise the subject's safety or adherence to the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Induction and maintenance Phase Efficacy- Crohn's Disease Activity Index (CDAI) | Week 12 and week 52
  Change from baseline in Crohn's Disease Activity Index (CDAI) score at Week 12 and Week 52 The CDAI total score ranges from 0 to over 600. Higher scores mean a worse outcome.
Maintenance Phase Efficacy - Simple Endoscopic Score for Crohn's disease (SES-CD) | Week 52
  Change from baseline in Simple Endoscopic Score for Crohn's disease (SES-CD) at Week 52
  The SES-CD is an endoscopic grading system that consists of a composite score based on 4 components: the size of mucosal ulcers, the extent of the ulcerated surface, the endoscopic extension, and the presence of stenosis (26). Each of the 4 SES-CD components are assessed in the 5 segments of the ileum and colon: ileum, right, transverse, left, and rectum. The SES-CD is the sum of the individual scores of each of the components across the 5 segments. The total score ranges from 0 to 60. Higher scores mean a worse outcome
Maintenance Phase Efficacy - Endoscopic response | Week 52
  Proportion of subjects with endoscopic response at Week 52
Maintenance Phase Efficacy - SES-CD ulcer subscore > 1 | Week 52
  Proportion of subjects with no SES-CD ulcer subscore > 1 in at least one segment at Week 52
Maintenance Phase Efficacy - CDAI clinical remission | Week 52
  Proportion of subjects with CDAI clinical remission at Week 52 Proportion of subjects with sustained CDAI clinical remission at Week 52
Maintenance Phase Efficacy - PRO-2 clinical remission | Week 52
  Proportion of subjects with patient reported outcome (PRO)-2 clinical remission at Week 52
Maintenance Phase Efficacy - CDAI clinical response | Week 52
  Proportion of subjects with CDAI clinical response (CDAI decrease from baseline ≥ 100 points) at Week 52
Maintenance Phase Efficacy - PRO-2 clinical response | Week 52
  Proportion of subjects with PRO-2 clinical response (≥ 30% decrease in average daily PRO-2 score (AP + SF) and both no higher than baseline) at Week 52
Maintenance Phase Efficacy - CDAI clinical response and endoscopic response | Week 52
  Proportion of subjects with CDAI clinical response and endoscopic response at Week 52
Maintenance Phase Efficacy - endoscopic remission | Week 52
  Proportion of subjects with endoscopic remission at Week 52
Extension Phase Safety- Adverse events | Weeks 64, 76, 88,100 and EOS
  Incidence of all treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and causally related TEAEs/SAEs Incidence of adverse events (AEs) leading to discontinuation
Extension Phase Safety - Hematology and coagulation | Weeks 64, 76, 88,100 and EOS
  Number of patients with clinically-significant abnormal laboratory parameters. Hematology: Hematocrit, hemoglobin, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, platelet count, red blood cells; white blood cells Coagulation: International normalized ratio, activated partial thromboplastin time, fibrinogen, prothrombin time
Extension Phase Safety - Biochemistry | Weeks 64, 76, 88,100 and EOS
  Number of patients with clinically-significant abnormal laboratory parameters. Albumin, total protein, aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), total bilirubin, gamma glutamyl transferase (GGT), lactate dehydrogenase (LDH), lipase, amylase, creatinine, creatinine clearance, urea, chloride, bicarbonate, sodium, potassium, calcium, phosphate, uric acid, glucose, total cholesterol, LDL cholesterol (direct), HDL cholesterol, triglycerides, creatine phosphokinase (CPK), high sensitivity troponin I and T, N-terminal prohormone of brain natriuretic peptide (NT-proBNP)

SECONDARY OUTCOMES:
Induction Phase Efficacy - SES-CD | Week 12
  Change from baseline in Simple Endoscopic Score for Crohn's disease (SES-CD) at Week 12
Induction Phase Efficacy - Endoscopic response | Week 12
  Proportion of subjects with endoscopic response at Week 12
Induction Phase Efficacy-SES-CD ulcer subscore > 1 | Week 12
  Proportion of subjects with no SES-CD ulcer subscore > 1 in at least one segment at Week 12
Induction Phase Efficacy-CDAI clinical remission | Week 12
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) clinical remission (CDAI score < 150) at Week 12 The total CDAI score ranges from 0 to over 600. Higher scores mean a worse outcome
Induction Phase Efficacy-PRO-2 clinical remission | Week 12
  Proportion of subjects with patient reported outcome (PRO)-2 clinical remission (Combination of average daily abdominal pain score ≤ 1.0 plus average daily soft or liquid stool frequency ≤ 2.8 and both no higher than baseline) at Week 12
Induction Phase Efficacy-CDAI clinical response | Week 12
  Proportion of subjects with CDAI clinical response (CDAI decrease from baseline ≥ 100 points) at Week 12 The total CDAI score ranges from 0 to over 600. Higher scores mean a worse outcome
Induction Phase Efficacy-PRO-2 clinical response | Week 12
  Proportion of subjects with PRO-2 clinical response at Week 12
Induction Phase Efficacy-CDAI clinical response and endoscopic response | Week 12
  Proportion of subjects with CDAI clinical response (CDAI decrease from baseline ≥ 100 points) and endoscopic response (Simple Endoscopic Score for Crohn's disease (SES-CD) decrease from baseline ≥ 50%) at Week 12
  The total CDAI score ranges from 0 to over 600. Higher scores mean a worse outcome The total SES-CD score ranges from 0 to 60. Higher scores mean a worse outcome.
Induction Phase Efficacy - endoscopic remission | Week 12
  Proportion of subjects with endoscopic remission at Week 12

CONTACTS AND LOCATIONS:
Locations (148):
- United States (43):
  - IMC Gulf Coast Gastroenterology, PC, Fairhope, Alabama
  - Scottsdale Gastroenterology Specialists, Scottsdale, Arizona
  - GI Alliance -Gurnee, Sun City, Arizona
  - Hoag Hospital, Irvine, California
  - United Medical Doctors, Murrieta, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Clinical Research Of Brandon, LLC, Brandon, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Auzmer Research, Lakeland, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Sarkis Clinical Trials - Parent, Ocala, Florida
  - Orlando Health, Inc., Orlando, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - Theia Clinical Research Centers, LLC, Temple Terrace, Florida
  - Northwestern University, Evanston, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Lucida Clinical Trials, LLC, New Bedford, Massachusetts
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - Henry Ford Columbus Center, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - OSU Inflammatory Bowel Disease Center, Hilliard, Ohio
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Rapid City Medical Center, LLC, Rapid City, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Novel Research, LLC, Bellaire, Texas
  - GI Alliance, Cedar Park, Texas
  - Baylor University Hospital, Dallas, Texas
  - GI Alliance - Garland, Garland, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - Houston Methodist Hospital, Houston, Texas
  - GI Alliance - Gurnee, Mansfield, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Richmond VA Medical Center, Richmond, Virginia
  - Gastroenterology Consultants of Southwest Virginia., Roanoke, Virginia
  - University of Washington, Seattle, Washington
- Belgium (6):
  - Hopital Universitaire de Bruxelles - Hopital Erasme, Brussels
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Wallonie Picarde, Tournai
  - CHU UCL Namur, Yvoir
- Czechia (6):
  - SurGal Clinic s.r.o., Brno
  - Vojenska nemocnice Brno, Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - PreventaMed s.r.o., Olomouc
  - ISCARE a.s., Prague
  - Nemocnice Slany, Slaný
- France (19):
  - CHU Amiens, Amiens
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Clermont Ferrand - Hopital d'Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon - Hôpital Bocage Central, Dijon
  - CHU de Grenoble - Hôpital Michallon, Grenoble
  - Centre Hospitalier Départemental Vendée - Les Oudairies, La Roche-sur-Yon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Lille - Hôpital Claude Huriez, Lille
  - Hôpital Nord - CHU Marseille, Marseille
  - Hopital Saint Eloi, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - Institut des MICI, Neuilly-sur-Seine
  - CHU Nice - Hôpital de l'Archet 2, Nice
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Hopital Rangueil, Toulouse
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (12):
  - Charite-Campus Benjamin Franklin Medizin.Klin.I, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Universitaetsklinikum Brandenburg an der Havel, Brandenburg
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main
  - Hamburgisches Forschungsinstitut fuer Chronisch Entzuendliche Darmerkrankungen, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - St. Marienkrankenhaus, Ludwigshafen
  - LMU - Campus Grosshadern, München
  - Universitaetsklinikum Ulm, Ulm
- Hungary (7):
  - Bekes Varmegyei Kozponti Korhaz, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Clinfan Szolgaltato Kft., Szekszárd
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Italy (9):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Ospedaliera Universitaria Renato Dulbecco di Catanzaro, Catanzaro
  - Ospedale San Raffaele, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Università Campus Bio-Medico di Roma, Roma
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Netherlands (5):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Radboud UMC, Nijmegen
  - ETZ Elisabeth, Tilburg
  - Bernhoven Uden, Uden
- Poland (22):
  - Centrum Medyczne Medis, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Santa Sp. z o.o. Sp. K Polimedica PTG Kielce, Kielce
  - Mz Badania Slowik Zymla Sp J, Knurów
  - Centrum Medyczne Plejady, Krakow
  - AMICARE spółka z ograniczoną odpowiedzialnością spółka komandytowa, Lodz
  - ALLMEDICA sp. z o. o., Nowy Targ
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - Trialmed CRS, Piotrkow Trybunalski
  - NSZOZ Termedica - Centrum Badan Klinicznych, Poznan
  - SOLUMED Centrum Medyczne, Poznan
  - Twoja Przychodnia PCM, Późna
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Kiepury Clinic MAŁGORZATA JARNOT SPECJALISTYCZNA PRAKTYKA GINEKOLOGICZNO-POŁOŻNICZA, Sosnowiec
  - DC-MED, Swidnica
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne Sp. z o. o., Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Medical Network Spolka z o.o, Warsaw
  - NZOZ VIVAMED Jadwiga Miecz, Warsaw
  - Melita Medical Sp. Z O. O., Wroclaw
  - ETG Zamosc, Zamość
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Lecznej, Łęczna
- Romania (5):
  - S.C Delta Health Care S.R.L, Bucharest
  - SC Centrul Medical Medicum SRL, Specialitatea Gastroenterologie, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - S.C Pelican Impex S.R.L, Oradea
  - Valahia Medical SRL, Ploieşti
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - Endomed, s.r.o., Košice
  - KM Management spol. s r.o., Nitra
  - Gastro I, s.r.o., Prešov
  - Penta hospitals SK, a.s., Rimavská Sobota
- Spain (8):
  - Centro Medico Teknon, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital General Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Clinica Gaias - Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia